CLINICAL TRIAL: NCT04872348
Title: An Observational Multicenter Clinical Study To Assess The Safety And Effectiveness Of The OMNI® Surgical System In Pseudophakic Eyes With Primary Open Angle Glaucoma (ORION 2.0)
Status: Completed | Type: Observational
Sponsor: Sight Sciences, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 07355
Record Dates: First submitted 2021-04-29; First posted 2021-05-04 (Actual); Results first posted 2025-05-11 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Glaucoma, Open-Angle
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Eyes receiving OMNI intervention after medication washout
  Interventions: Device: OMNI® Surgical System
- Eyes receiving OMNI intervention without medication washout
  Interventions: Device: OMNI® Surgical System

INTERVENTIONS:
Device: OMNI® Surgical System — The OMNI® Surgical System is indicated for canaloplasty (microcatheterization and transluminal viscodilation of Schlemm's canal) followed by trabeculotomy (cutting of trabecular meshwork) to reduce intraocular pressure in adult patients with primary open-angle glaucoma.

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of the OMNI® Surgical System in subjects who have undergone canaloplasty and trabeculotomy using OMNI® Surgical System without any concomitant surgery in pseudophakic eyes with mild to moderate primary open angle glaucoma (POAG) at least 150 days prior to enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Treated with OMNI® Surgical System as a standalone procedure in pseudophakic eye with mild to moderate primary open angle glaucoma at least 150 days prior to enrollment.

Exclusion Criteria:

* Systemic disease that, in the opinion of the Investigator, would put the subject's health at risk and/or prevent completion of required study visits.
* Ocular pathology which, in the Investigator's judgment, would either place the subject at increased risk of complications or contraindicate washout, place the subject at risk of significant vision loss during the study period or interfere with compliance to elements of the study protocol (e.g., returning to Investigator's office for follow-up visits).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects treated with OMNI® Surgical System as a standalone procedure in pseudophakic eye with mild to moderate primary open angle glaucoma
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-11-02 (Actual); Study Completion 2023-11-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Eye Specialists of Georgia, Atlanta, Georgia
  - Grene Vision Group, Wichita, Kansas
  - Minnesota Eye Consultants, Bloomington, Minnesota
  - Northern New Jersey Eye Institute, Orange, New Jersey
  - Oklahoma Eye Surgeons, Oklahoma City, Oklahoma
  - University Eye Specialists, Maryville, Tennessee
  - El Paso Eye Surgeons, El Paso, Texas
  - Ophthalmology Associates - Fort Worth, Fort Worth, Texas
  - Utah Eye Centers, Ogden, Utah
  - Virginia Eye Consultants, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Washout: Eyes receiving OMNI intervention after medication washout.
- No Washout: Eyes receiving OMNI intervention without medication washout
Period: Overall Study
Arm/Group | Washout | No Washout
Started | 18 | 10
Completed | 18 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Washout | No Washout | Total
Number analyzed (Participants) | 18 | 10 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.0 (8.2) | 76.0 (4.7) | 75.4 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 7 | 18
  Male | 7 | 3 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 0 | 6
  Not Hispanic or Latino | 11 | 10 | 21
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 5 | 6
  White | 17 | 4 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 18 | 10 | 28

OUTCOME MEASURES:

1. Primary Outcome: Change in Intraocular Pressure (IOP)
Description: Percent change in unmedicated diurnal intraocular pressure (DIOP/washout) or medicated intraocular pressure (IOP/no washout) compared to baseline.
Time Frame: 18 months
Population: Intent To Treat
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Washout | No Washout
Number analyzed (Participants) | 13 | 8
percent change | 38.2 (15.53) | 30.1 (24.14)

2. Primary Outcome: Change in Number of Medications
Description: Mean change in the number of ocular hypotensive medications compared to baseline.
Time Frame: 18 months
Population: Intent To Treat
Measure: Mean (Standard Deviation); unit: number of medications
Arm/Group | Washout | No Washout
Number analyzed (Participants) | 15 | 8
number of medications | -1.13 (1.06) | -0.13 (1.25)

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Washout | No Washout
All-Cause Mortality (participants affected / at risk) | 0/18 | 1/10
Serious Adverse Events (participants affected / at risk) | 0/18 | 1/10
Other Adverse Events (participants affected / at risk) | 12/18 | 7/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Washout (N=18) | No Washout (N=10)
Death (General disorders) | 0 (0) | 1 (1) — Cause unknown
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Washout (N=18) | No Washout (N=10)
IOP increase above baseline at 1mont or greater (Eye disorders) | 1 (1) | 1 (2) — IOP increase >=10 mmHg above baseline IOP at >=1 month visit
Layered Hyphema (Eye disorders) | 0 (0) | 1 (1)
Secondary Surgical Intervention (Eye disorders) | 1 (1) | 0 (0)
Corneal edema after 1 week (Eye disorders) | 0 (0) | 1 (1)
IOL dislocation and/or damage (Eye disorders) | 0 (0) | 1 (1)
Posterior capsular opacification (Eye disorders) | 1 (1) | 2 (2)
Iridodialysis or significant iris damage (Eye disorders) | 0 (0) | 1 (1)
Conjunctival hyperemia (Eye disorders) | 1 (1) | 0 (0)
Corneal epithelial microcysts (Eye disorders) | 0 (0) | 1 (1)
Dizziness (General disorders) | 0 (0) | 1 (1)
Dry Eye (General disorders) | 2 (2) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 0 (0) | 1 (1)
Headache (General disorders) | 0 (0) | 1 (1)
Intraocular pressure increased (Eye disorders) | 0 (0) | 1 (1)
Iridocele (Eye disorders) | 1 (1) | 0 (0)
Iris adhesions (Eye disorders) | 1 (1) | 0 (0)
Iris atrophy (Eye disorders) | 1 (1) | 0 (0)
Iris transillumination defect (Eye disorders) | 3 (3) | 0 (0)
Nausea (General disorders) | 0 (0) | 1 (1)
Pigment dispersion syndrome (Eye disorders) | 2 (2) | 0 (0)
Punctate keratitis (Eye disorders) | 1 (1) | 0 (0)
Pupillary reflex impaired (Eye disorders) | 0 (0) | 1 (1)
Retinal drusen (Eye disorders) | 1 (1) | 0 (0)
Sinus pain (General disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After Sponsor's publication of trial results, the Institution and Principal Investigator may publish the results of the Study generated by the Institution, subject to the obligations of the CTA, and prior approval of Sponsor in writing. The Institution shall furnish Sponsor with a written copy of any proposed publication or disclosure at least 60 days prior to submission for publication or disclosure. Sponsor may request changes or other measures to ensure the information is fairly stated.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-30): https://cdn.clinicaltrials.gov/large-docs/48/NCT04872348/Prot_SAP_000.pdf